CLINICAL TRIAL: NCT04079699
Title: Predicting Prostate Cancer Using a Panel of Plasma and Urine Biomarkers Combined in an Algorithm in Elderly Men Above 70 Years
Brief Title: Predicting Prostate Cancer in Elderly Men
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Odense University Hospital (Other)
Responsible Party: Principal Investigator, Mads Hvid Poulsen, MD, PhD, Associate professor, Odense University Hospital
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Diagnostic
Other Study IDs: DaProCa4
Record Dates: First submitted 2019-09-03; First posted 2019-09-06 (Actual); Last update posted 2019-09-06 (Actual); Status verified 2019-09

CONDITIONS: Prostate Cancer (Diagnosis)
MeSH Terms: conditions — Prostatic Neoplasms; Disease | interventions — Liquid Biopsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Liquid Biopsy (Experimental): Experimental arm where the "liquid biopsy" decides whether to perform an prostate biopsy or not
  Interventions: Diagnostic Test: Liquid Biopsy
- Standard Biopsy (Other): Standard arm, where every patient receives a standard prostate biopsy
  Interventions: Diagnostic Test: Standard biopsy

INTERVENTIONS:
Diagnostic Test: Liquid Biopsy — Measuring biomarkers in blood and urine samples
  Arms: Liquid Biopsy
Diagnostic Test: Standard biopsy — Histological examination of tissue biopsies
  Arms: Standard Biopsy

SUMMARY:
We aim to analyze whether the "liquid biopsy" model could increase the specificity of detecting men with an aggressive (defined as Gleason score ≥ 7) prostate cancer and thereby reduce the proportion of men who undergo prostate biopsy, while at the same time maintaining the same sensitivity to detect aggressive prostate cancer as the PSA test alone. Using blood and urine biomarkers together with an algorithm, which incorporates the clinical data, we aim to identify patients who have a high risk of having an aggressive prostate cancer. By performing this non-invasive test we expect that we can reduce need for prostate biopsy and reduce the detection of patients with an indolent prostate cancer (defined by Gleason score ≤ 6). Thereby we aim to reduce the side effects of transrectal ultrasound guided biopsy of the prostate and side-effects of living with an indolent cancer.

DETAILED DESCRIPTION:
BACKGROUND Prostate biopsy is currently the standard of care for prostate cancer diagnosis, oftentimes reflexed after the detection of an elevated serum prostate-specific antigen (PSA). Unfortunately, prostate biopsy is not without potential complications, which include discomfort, pain, bleeding, and infections ranging from cystitis to septic sepsis and even death. Bleeding has been reported in 6-13% of patients undergoing prostate biopsy, while 0.3-4% experience admission with sepsis. Furthermore, some newly diagnosed prostate cancers are indolent while other may be more aggressive with metastatic potential, with resultant risk of death. A PSA level ≥4.0 ng/ml is frequently used as a threshold warranting a biopsy evaluation. Elevated PSA level may reflect benign prostatic hyperplasia (BPH), inflammation, or malignancy. Some series suggest that only 20-30% of patients with PSA 4 - 10 ng/ml, have prostate cancer, resulting in a high number of patients undergoing an unnecessary biopsy. We recently reported the ability of "Liquid Biopsy" to predict the presence of aggressive prostate cancer using a combination of biomarkers detected in urine and peripheral blood plasma. Concluding that "Liquid Biopsy" can predict the presence of aggressive prostate cancer (GS ≥7).

AIM With this study we want of compare "Liquid Biopsy", defined by our blood and urine panel against prostate biopsy in a large-scale randomized manner including men referred for a biopsy due to the suspicion of prostate cancer over the age of 70 (elderly).

OBJECTIVE The primary objectives of this study are to test the ability of the "liquid biopsy" to

1. Detect as many patients with aggressive prostate cancer as the standard method (PSA).
2. Reduce the number of prostate biopsy sets taken and thereby reduce the number of patients detected with indolent prostate cancer.

The secondary objectives are to evaluate

1. The economic effect of implementation of the test with regard to reduced biopsies taken, iatrogenic infectious disease and reduced control of indolent prostate cancer.
2. The association of the liquid biopsy to tumor grade and tumor volume in biopsied men.
3. The Quality of life.
4. Progression and survival: overall survival, prostate cancer specific survival, PSA recurrence, time to metastases, time to castration resistance
5. Safety

ELIGIBILITY:
Inclusion Criteria:

* Suspicion of prostate cancer due to elevated PSA, and/or palpable tumor in the prostate
* Indication for digital rectal examination and trans-rectal ultrasound with biopsy
* Age: 70 years or above
* PSA: 20 or above
* Able to provide informed written consent (competent adults only)

Exclusion Criteria:

* Previously diagnosed with prostate cancer
* Receiving treatment influencing PSA levels
* Medical conditions that may interfere with the study such as previously cancer-related therapy
* Life expectancy of less than 10 years
* MRI of the prostate within the last 2 years
* Digital rectal examination of the prostate within 24 hours or ejaculation within 24 hours

Min Age: 70 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Older Adult
Gender Based: Yes — We can only include persons born with a prostate.
Enrollment: 700 (Estimated)
Dates: Start 2019-10-01 (Estimated); Primary Completion 2039-10-01 (Estimated); Study Completion 2039-10-01 (Estimated)

PRIMARY OUTCOMES:
Test sensitivity | 2 years
  Number of detected patients with aggressive prostate cancer, defined as Gleason score ≥ 7.
Test specificity | 20 years
  Number of patients who had prostate biopsies

CONTACTS AND LOCATIONS:
Overall Officials: Lars Lund, MD, DMSci, Study Director — Odense University Hospital

IPD SHARING:
Plan to Share IPD: No
Personal data is maintained in a safe database with logging and only anonymized data will be shared if needed.